CLINICAL TRIAL: NCT01777412
Title: An Open-label Phase 1b Study of Avastin® (Bevacizumab) for the Treatment of Acute Optic Neuritis and/or Transverse Myelitis in Neuromyelitis Optica (NMO) and Neuromyelitis Optica Spectrum Disorder (NMOSD).
Brief Title: Efficacy of Bevacizumab (Avastin) in Treatment of Acute NMO Exacerbations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry); Guthy Jackson Charitable Foundation (Other)
Responsible Party: Principal Investigator, Michael Levy, Assistant Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Avastin_NMO_1
Record Dates: First submitted 2013-01-21; First posted 2013-01-28 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Neuromyelitis Optica; Neuromyelitis Optica Spectrum Disorder
Keywords: NMO; NMOSD; NMO-IgG; Aquaporin-4; AQP4; anti-AQP4
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental): Bevacizumab 10 mg/kg intravenous infusion at onset of exacerbation and, if needed, a second time during the plasma exchange phase.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin

SUMMARY:
This is a phase 1b interventional trial of bevacizumab (Avastin®) to evaluate the tolerability/safety and preliminary efficacy of bevacizumab (Avastin®) as add-on therapy for treatment of acute optic neuritis and/or transverse myelitis in neuromyelitis optica (NMO) and neuromyelitis optica spectrum disorder (NMOSD). A single infusion of Avastin® is added to standard-of-care high dose steroids and an additional dose of Avastin® is added to plasma exchange (if necessary). The primary outcomes are clinical changes in the Expanded Disability Severity Scale, Timed 25-foot Walk and Low Contrast Visual Acuity, MRI parameters and safety.

DETAILED DESCRIPTION:
Study Objective: The overall objective is to evaluate the tolerability/safety and efficacy of adding bevacizumab (Avastin®) to standard of care therapy in improving clinical and radiologic outcomes of acute optic neuritis and/or transverse myelitis in neuromyelitis optica and neuromyelitis optica spectrum disorders.

Primary Objective: To compare the clinical and radiographic outcome following acute optic neuritis and/or transverse myelitis in NMO/NMOSD in patients who receive 1-2 doses of 10 mg/kg dose of bevacizumab (Avastin®) in addition to standard medical therapy.

Secondary Objectives:

* To determine the effect of Avastin on NMO clinical scores (Expanded Disability Status Scale, Timed 25-foot Walk and Low Contrast Visual Acuity [LCVA]).
* To evaluate the safety and tolerability of a 10 mg/kg dose of intravenous Avastin.
* To determine the frequency of adverse events with Avastin in this patient population.
* To determine the effect of Avastin on MRI lesion size and extent.

The duration of the investigation is 1-2 years.

ELIGIBILITY:
Subjects eligible for enrollment must meet all of the following criteria:

1. Able and willing to provide written informed consent.
2. 18-70 years of age.
3. New acute optic neuritis and/or transverse myelitis. A clinical event is defined as an episode of inflammation in the spinal cord and/or optic nerve leading to neurologic symptoms not ascribed to another disease process.
4. Known or suspected diagnosis of NMO according to the 2006 revisions of the Wingerchuk diagnostic criteria for NMO or AQP4 positive NMOSD per the EFNS Guidelines. For NMO, subjects must have two absolute criteria:

   1. optic neuritis
   2. myelitis and at least two of three supportive criteria:
   3. presence of a contiguous spinal cord MRI lesion extending over three or more vertebral segments,
   4. MRI criteria NOT satisfying the revised McDonald diagnostic criteria for MS [Polman, 2011]
   5. NMO-IgG (AQP4) in serum. For NMOSD, subjects must have longitudinally extensive transverse myelitis (LETM) recurrent isolated optic neuritis (RION)/bilateral optic neuritis (BON), or opticospinal multiple sclerosis (OSMS) that is AQP4 antibody positive
5. A female subject is eligible to enter the study if she is:

A. Not pregnant or nursing; B. Of non-childbearing potential (i.e. women who have had a hysterectomy, are postmenopausal, which is defined as >2 years without menses (female subjects who have been post-menopausal for <2 years must be confirmed with Follicle Stimulating Hormone (FSH) and estradiol levels), have both ovaries surgically removed or have current documented tubal ligation); or,

C. Of childbearing potential (i.e. women with functional ovaries and no documented impairment of oviductal or uterine function that would cause sterility). This category includes women with oligomenorrhoea (even severe), women who are perimenopausal or have just begun to menstruate. The subject must have a negative serum pregnancy test at screening and agrees to one of the following:

i. Complete abstinence from intercourse for the period from consent into the study until 6 months after the last dose of investigational product; or, ii. Consistent and correct use of one of the following acceptable methods of birth control for the period from consent into the study until 6 months after the last dose of investigational product:

1. Oral contraceptives (either combined or progesterone only)
2. Injectable progesterone
3. Levonorgestrel implants
4. Estrogenic vaginal ring
5. Percutaneous contraceptive patches
6. Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of <1% per year
7. Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study; this male must be the sole partner for the subject
8. Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository).

Subjects meeting any of the following criteria are not eligible and cannot enroll in the study:

1. Evidence or history of clinically significant infection including:

   1. Chronic or ongoing active infectious disease requiring long term systemic treatment such as, but not limited to: PML, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis, or active hepatitis C.
   2. Positive test for HBsAg.
   3. Prior history, or suspicion, of tuberculosis (TB)
   4. History of positive serology for HIV.
2. Past or current malignancy, except for

   1. Cervical carcinoma Stage 1B or less
   2. Non-invasive basal cell and squamous cell skin carcinoma
   3. Cancer diagnoses with a duration of complete response (remission) >5 years
   4. A history of hematologic malignancy excludes a subject from participation, regardless of response.
3. Recent major surgery within the last 28 days.
4. Significant concurrent, uncontrolled medical condition including, but not limited to, cardiac, renal, hepatic, hematological, gastrointestinal, endocrine, immunodeficiency syndrome, pulmonary, cerebral, psychiatric, or neurological disease which could affect the subject's safety, impair the subject's reliable participation in the trial, impair the evaluation of endpoints, or necessitate the use of medication not allowed by the protocol.
5. Use of an investigational drug or other experimental therapy for a condition other than NMO within 4 weeks, 5 pharmacokinetic half lives or duration of biological effect (whichever is longer) prior to screening.
6. Current participation in any other interventional clinical trial. Participation in non-interventional trial requires approval of the protocol by investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levy, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- See also: Johns Hopkins NMO Clinic — http://www.hopkinsmedicine.org/neurology_neurosurgery/research/neuromyelitis-optica-research-lab/nmo-clinic.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Bevacizumab 10 mg/kg intravenous infusion at onset of exacerbation and, if needed, a second time during the plasma exchange phase in additional 5 days of 1000 mg methylprednisolone infusion. There was no placebo or comparator group.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (15.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Diagnosis [Number; unit: participants]
  NMO/NMOSD | 7
  High risk for NMO | 3
Anti-AQP4 antibody serostatus [Number; unit: participants]
  Positive | 6
  Negative | 4

OUTCOME MEASURES:

1. Primary Outcome: Baseline Expanded Disability Status Score (EDSS)
Description: EDSS
  The EDSS provides a total score on a scale that ranges from 0 to 10. The first levels 1.0 to 4.5 refer to people with a high degree of ambulatory ability and the subsequent levels 5.0 to 9.5 refer to the loss of ambulatory ability.
Time Frame: Admission to hospital
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bevacizumab
Number analyzed (Participants) | 10
units on a scale | 3.5 [2.0 to 7.0]

2. Primary Outcome: Safety Assessment and Side Effects
Description: Frequency and severity of adverse events and side effects. Serious adverse events are considered those which are life threatening, lead to hospitalization and related to the drug. Side effects are considered minor effects of the experimental drug that do not significantly impact the care of the patient with the experimental drug.
Time Frame: 91 days
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 10
participants
  Serious Adverse Event: Hospitalization | 1
  Side Effects | 0

3. Primary Outcome: Follow-Up Expanded Disability Status Score (EDSS)
Description: as for outcome 1
Time Frame: Follow-up visit 91 days after admission
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Bevacizumab
Number analyzed (Participants) | 10
units on a scale | 3.0 [1.75 to 6.5]

ADVERSE EVENTS:
Time Frame: 91 days
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=10)
Hospitalization for Urinary Tract Infection (Infections and infestations) | 1 (1) — 47 days after infusion of bevacizumab, patient developed a urinary tract infection that required hospitalization for 1 night and initiation of antibiotics. The infection was treated completely without complications.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=10)
Headache (Nervous system disorders) | 1 (1) — Headache during the infusion of bevacizumab was noted. The headache resolved with fluids.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No